CLINICAL TRIAL: NCT01203657
Title: Tai Chi, Vitality and Activity in a Community Setting
Brief Title: UCLA Tai Chi in a Community Setting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: UCLA-TCC01
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Physical Activity; Fatigue
Keywords: exercise; physical activity; tai chi
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Tai Ji; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): Tai Chi instruction, 2x week in a community senior center setting
  Interventions: Behavioral: Tai Chi
- Wait List Control (No Intervention): This is a wait list control group. There is no active or placebo intervention.

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi classes, 60 minutes, 2x week
  Other Names: exercise; relaxation
  Arms: Tai Chi

SUMMARY:
Although a number of studies have examined the effects of Tai Chi in older adult populations, few have methodically assessed its effects on vitality, fatigue and physical activity. Some studies have shown that fatigue relates to negative mood and poor health-related quality of life in older persons.

Tai Chi is an ancient Chinese form of calisthenics that utilizes the body's internal energy (chi), mind, and breathing; which may be a useful exercise for older adults in increasing their activity level. A twenty-four of Yang style of Tai Chi is a simple form of Tai Chi that is particularly well-suited for older adults. This proposed study to investigate the effects of a Tai Chi intervention on decreasing fatigue level, and increasing level of activity in healthy older adults.

The investigators research group has focused on the Tai Chi as a strategy to reduce stress and improve sleep, and their preliminary evidence suggest it strongly affects energy level and vitality. The investigators are focused on taking this intervention into the community testing its efficacy. The investigators preliminary data shows that Tai Chi is of benefit to older adults; however, this study will test whether their research findings are generalizable to community settings.

Tai Chi-naïve participants from Culver City Senior Center will receive a 10-week Tai Chi. The investigators will compare this group to a wait-list control group. All subjects will receive a packet of questionnaires of pre- and post-intervention vitality, fatigue and health-related quality of life. Subjects will also be given an activity monitor to wear for 2 days before they start the Tai Chi class and for 2 days after they complete the class, to determine if there is a change in general physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Older adult > 60 years of age

Exclusion Criteria:

* Older adults who have severe osteoarthritis or chronic pain disorders
* Non ambulatory
* Any condition that would adversely impact their participation in Tai Chi

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Immediately post-intervention (10 weeks)
  Objectively assessed physical activity measured using accelerometers

SECONDARY OUTCOMES:
Vitality | Immediately post-intervention (10 weeks)
  Measures of fatigue, mood, perceived stress and vitality, administered via self-report

CONTACTS AND LOCATIONS:
Overall Officials: Sarosh Motivala, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States